CLINICAL TRIAL: NCT02640898
Title: Docetaxel-based Chemoradiotherapy Plus Periradiation Chemotherapy in R0 Gastric Cancer
Brief Title: Docetaxel-based Chemoradiotherapy Plus Periradiation Chemotherapy Compared With INT 0116 Adjuvant Arm in Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, Docetaxel-based chemoradiotherapy plus periradiation chemotherapy in R0 gastric cancer, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGH201510
Record Dates: First submitted 2015-12-19; First posted 2015-12-29 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FU-based chemoradiotherapy (Active Comparator): patients will be treated with the INT0116 regimen.
  Interventions: Radiation: FU-based chemoradiotherapy
- docetaxel-based chemoradiotherapy (Experimental): patients will be treated with modified DCF chemotherapy in combination with docetaxel-based chemoradiotherapy.
  Interventions: Radiation: docetaxel-based chemoradiotherapy

INTERVENTIONS:
Radiation: docetaxel-based chemoradiotherapy — experimental:Patients with Zubrod performance status (PS) of 0-2 received up to 2 21-day cycles of pre- and post-radiation chemotherapy (docetaxel 37.5 mg/m2 on days 1 and 8, cisplatin 25 mg/m2 on days 1-3, and a continuous infusion of fluorouracil (FU) 750 mg/m2 on days 1-5), respectively. CCRT between pre- and post-radiation chemotherapy was initiated on day 43 and consisted of 3-dimensional conformal intensity-modulated radiation therapy (45 Gy) plus concurrent docetaxel 20 mg/m2 weekly for 6 weeks;
  Other Names: a docetaxel arm
  Arms: docetaxel-based chemoradiotherapy
Radiation: FU-based chemoradiotherapy — The adjuvant treatment consisted of 425mg/m2 of bolus fluorouracil(5-FU) per day, 20 mg/m2 of leucovorin (LV), per day, for 5 days, followed by 45Gy of radiation with current 5-FU ( 400mg/m2 ) and LV (20mg/m2) as an intravenous bolus on each of of the first four days and the last three days of irradiation. One month after the completion of radiotherapy, two 5-day cycles of 5-FU and FV chemotherapy were given one month apart.
  Other Names: the INT 0116 adjuvant arm
  Arms: FU-based chemoradiotherapy

SUMMARY:
Although the intergroup 0116 trial was the first to demonstrate that adjuvant chemoradiotherapy offers a significant survival benefit in completely resected gastric cancer,it is more toxic and less effective. It is reasonable to optimize this regimen.

DETAILED DESCRIPTION:
The intergroup 0116 trial was the first to demonstrate that adjuvant chemoradiotherapy offers a significant survival benefit. In this study, 556 patients with R0 resected gastric cancer were randomly assigned to surgery plus postoperative chemoradiotherapy or to surgery alone. The adjuvant treatment consisted of 425 mg per square meter of bolus fluorouracil per day, 20 mg per square meter of leucovorin , per day, for 5 days, followed by 45 Gy of radiation with current fluorouracil ( 400mg per square meter ) and leucovorin (20mg per square meter) as an intravenous bolus on each of of the first four days and the last three days of irradiation. One month after the completion of radiotherapy, two 5-day cycles of fluorouracil and leucovorin chemotherapy were given one month apart. Patients in the adjuvant arm achieved a significant 3-year overall and relapse-free survival benefit of 9% and 17%, respectively.

Despite the improvement in outcome, up to 120 of 281 patients in the chemoradiotherapy arm relapsed in local regional or/and distant sites within 3 years of potentially curative resection. Notably, the patients receiving chemoradiotherapy had a higher rate of distant metastasis compared with the control arm (40/281 vs 32/275), indicating that bolus 5-FU/LV was not suboptimal to control the development of distant metastases. Furthermore, the toxicity in INT 0116 trial was substantial, with grade 3 or higher overall toxicities observed in 73% of the cases. As a result, only 64% of the patients were able to complete protocol therapy. Obviously, it is reasonable to optimize the Intergroup 0116 chemoradiotherapy regimen.

Docetaxel, as a monotherapy, is active in both first- and second-line treatment of advanced stage gastric cancer. In addition, in vitro and in vivo studies have demonstrated that docetaxel is a potent radiosensitizer in human cancer cell lines, making it an attractive agent combined with radiation. A phase I study has identified the phase II recommended dose of docetaxel as 20mg/m2 weekly for six weeks when administered with concurrent chest radiation of 60 Gy.

Furthermore, docetaxel when added to standard cisplatin and infused fluorouracil (DCF regimen) demonstrated an advantage in survival, time to progression, and response rate (RR) over cisplatin and fluorouracil (CF) in a randomized phase Ⅲ trial, but the toxicity profile associated with the DCF regimen was significant. In addition, a favorable RR and median overall survival for DCF over epirubicin, cisplatin, protracted venous infusion fluorouracil (ECF) has been seen in a randomized phase Ⅱ trial.

Two large phase III trials has demonstrated that the addition of perioperative chemotherapy (ECF) or adjuvant chemotherapy (S1) to radical surgery could significantly improve surgical outcomes in localized gastric cancer as compared with surgery alone in terms of progression-free and overall survival. These results suggest that adjuvant and neoadjuvant chemotherapy may have excellent effects on both the primary tumor and micrometasatsis.

Based on these important findings, we designed a phase 3 trial to compared our novel docetaxel-based chemoradiotherapy regimen with the Intergroup 0116 adjuvant arm in patients with curatively resected gastric cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with microscopically confirmed stages IB through IIIB adenocarcinoma of the stomach or gastroesophageal junction, who underwent a potentially curative resection (ie, R0 resection);
* Zubrod performance status 0 to 1;
* No prior chemotherapy or prior radiation therapy to the treatment field;
* Age 20-75;
* Absolute granulocyte count (AGC) ≥2 × 109 cells/L, platelets ≥ 100× 109 cells/L, hemoglobin ≥ 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is acceptable)
* Adequate renal and hepatic function (serum creatinine ≤1.5 × upper limit of normal [ULN], bilirubin and AST ≤1.5 × ULN).

Exclusion Criteria:

* A history of prior upper abdominal radiotherapy or chemotherapy;
* Evidence of metastatic disease to distant organs, peritoneal carcinoma by computed tomography or positive cytology of peritoneal effusion;
* Prior malignancies (except cured cervical carcinoma in situ, non-melanoma skin cancer, or other curatively treated cancer with no evidence of disease for ≥5 years);
* active inflammatory bowel disease;
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
* Transmural myocardial infarction within the last 6 months;
* uncontrolled hypertension;
* Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 60 days before registration;
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
* Patients with Acquired Immune Deficiency Syndrome were excluded from the study because the treatments involved in this protocol may be significantly immunosuppressive.
* Hypersensitivity reaction to docetaxel;
* Uncontrolled neuropathy grade 2 or greater regardless of cause;
* Conditions precluding medical follow-up and protocol compliance;
* Pregnant or lactating women are excluded from study entry due to the embryotoxic effects of the protocol treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-12; Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | 3-year (36-month)
  survival time was measured from the date of study enrollment to the date of death or last follow-up

SECONDARY OUTCOMES:
progression free survival rate | 3-year (36-month)
  progression free survival was measured from the date of study entry to the first event (ie,local-regional relapse or progression, distant recurrence, or death of any cause)

CONTACTS AND LOCATIONS:
Overall Officials: tingfeng chen, MD, Principal Investigator — the ethic committee of shanghai genernal hospital
Locations (1):
- the Ethic Committee of Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Sulkes A, Smyth J, Sessa C, Dirix LY, Vermorken JB, Kaye S, Wanders J, Franklin H, LeBail N, Verweij J. Docetaxel (Taxotere) in advanced gastric cancer: results of a phase II clinical trial. EORTC Early Clinical Trials Group. Br J Cancer. 1994 Aug;70(2):380-3. doi: 10.1038/bjc.1994.310. PMID 7914428
- [Background] Choy H, Rodriguez FF, Koester S, Hilsenbeck S, Von Hoff DD. Investigation of taxol as a potential radiation sensitizer. Cancer. 1993 Jun 1;71(11):3774-8. doi: 10.1002/1097-0142(19930601)71:113.0.co;2-0. PMID 8098270
- [Background] Mauer AM, Masters GA, Haraf DJ, Hoffman PC, Watson SM, Golomb HM, Vokes EE. Phase I study of docetaxel with concomitant thoracic radiation therapy. J Clin Oncol. 1998 Jan;16(1):159-64. doi: 10.1200/JCO.1998.16.1.159. PMID 9440738
- [Background] Van Cutsem E, Moiseyenko VM, Tjulandin S, Majlis A, Constenla M, Boni C, Rodrigues A, Fodor M, Chao Y, Voznyi E, Risse ML, Ajani JA; V325 Study Group. Phase III study of docetaxel and cisplatin plus fluorouracil compared with cisplatin and fluorouracil as first-line therapy for advanced gastric cancer: a report of the V325 Study Group. J Clin Oncol. 2006 Nov 1;24(31):4991-7. doi: 10.1200/JCO.2006.06.8429. PMID 17075117